CLINICAL TRIAL: NCT04142190
Title: Influence of Corifollitropin Alfa (Elonva) on Embryo Morphokinetics and Fertility Treatment Outcome
Brief Title: Corifollitropin Alfa and Embryo Morphokinetics
Status: Completed | Type: Observational
Sponsor: Kinderwunsch Institut GmbH (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: FRED001
Record Dates: First submitted 2019-10-14; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Infertility
Keywords: follicle-stimulating hormone; embryo morphokinetics; reproductive medicine
MeSH Terms: conditions — Infertility | interventions — follitropin beta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ELONVA: Patients stimulated with Elonva
  Interventions: Drug: ELONVA
- PUREGON: Patients stimulated with Puregon
  Interventions: Drug: PUREGON

INTERVENTIONS:
Drug: ELONVA — Elonva is a solution for injection that contains the active substance corifollitropin alfa. It is available as a pre-filled syringe (100 and 150 micrograms).Elonva is used in women who are undergoing fertility treatment to stimulate the development of more than one mature egg at a time in the ovaries.
  Groups: ELONVA
Drug: PUREGON — Puregon contains the active substance follitropin beta. fertilisation). Puregon is administered to stimulate the ovaries to produce more than one egg at a time
  Groups: PUREGON

SUMMARY:
The study evaluates the influence of corifollitropin alfa (Elonva) on embryo morphokinetics and fertility treatment outcome in comparison to a control group stimulated with Follitropin beta (Puregon).

DETAILED DESCRIPTION:
Morphokinetic parameters of embryo development have been intensively investigated. However, little attention has been paid to the influence of ovarian stimulation on morphokinetic parameters. Gryshenko et al. found a significant difference in the fourth cell division time (t5) of embryos obtained after controlled ovarian hyperstimulation in long GnRH agonists and GnRH antagonist protocols. Furthermore, higher gonadotropin doses were found to slow down the development of the embryos.

Hence, the aim of this study is to investigate the influence of corifollitropin alfa (Elonva) on embryo morphokinetics and fertility treatment outcome in comparison to a control group stimulated with Follitropin beta (Puregon). The investigators hypothesize that there are differences in morphokinetic behavior of embryos within the different stimulation protocols.

A total of 742 embryos from 215 different patients suffering from infertility undergoing ovarian stimulation with Elonva and a total of 5148 embryos from 1136 patients undergoing ovarian stimulation with Puregon will be retrospectively analyzed. To exclude environmental factors the evaluation will distinguish between embryos cultured under 21% oxygen and embryos with reduced oxygen conditions (5% oxygen) in the embryoscope. Groups will be age and BMI matched.

All women included in the study underwent GnRH (Gonadotropin-releasing hormone) antagonist protocol controlled ovarian hyperstimulation. Patients received recombinant human follicle-stimulating hormone (Elonva; MSD Sharp &Dohme GMBH, Puregon; MSD Sharp & Dohme GMBH). ELONVA was administered for 7 days with subsequent administration of Puregon (MSD Sharp & Dohme GMBH) in case of further need of stimulation. Puregon was administered for 8-10 days with dosage adaption according to age, weight, serum anti-mullerian hormone (sAMH) concentration, and hormonal status. Trans-vaginal sonography was performed after 5 days of stimulation, followed by every second day until the day of oocyte retrieval. Ultrasonographical measurement was performed using a RIC 5-9-D 4D intravaginal probe of a GE Voluson E8 BT09 ultrasound machine (both from GE Healthcare Austria GmbH). GnRH antagonist (Cetrotide, Merck KGaA) was injected to avoid premature ovulation. Triggering was initiated 35 h before oocyte retrieval, administered with 5000-10,000 IU human chorionic gonadotropin (hCG) subcutaneously (Pregnyl, N.V. Organon), with dosage adaption according to body weight of the patient.

Follicles larger than 10 mm in diameter were aspirated under sedation (Propofol, Fresenius Kabi Austria GmbH; Rapifen, Janssen-Cilag Pharma GmbH) and transvaginal ultrasound guidance (GE Healthcare Austria GmbH). Follicular fluid (FF) were examined for oocytes under constant conditions of 37 °C in an IVF workstation L24E with heating stage (K-SYSTEMS Kivex Biotec A/S). Intracytoplasmic sperm injection (ICSI) was performed on all metaphase II (MII) oocytes 4-5h after oocyte retrieval according to our standard operating procedure in both groups of patients.

After oocyte retrieval and fertilization, oocytes were cultivated in universal culture medium (Gynemed Medizinprodukte GmbH & Co. KG, Germany). After 14-16 h, fertilization check was performed. All normal fertilized embryos with two pronuclei (PN) were then cultured using Embryoslide dishes in Embryoscope® time-lapse incubator (both Vitrolife AB, Sweden). With the built-in camera and microscope, images of the developing embryo were taken every 15 min in seven different layers. Definition of morphokinetic parameters was performed according to the criteria proposed by Ciray et al. and was analyzed with software developed for time-lapse image analysis (Embryoviewer® software; Vitrolife AB, Sweden).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-42
* BMI: 19-29.9
* Primary or secondary infertility
* Ovarian stimulation with Elonva/Puregon
* Embryos cultured in embryoscope

Exclusion Criteria:

* unexpected low response
* genetic testing

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Women suffering from infertility
Sampling Method: Probability Sample
Enrollment: 1351 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Time of pronuclei disappearance | 16-18 hours after fertilization
  Time of pronuclei disappearance in embryos of patients stimulated with ELONVA versus embryos of patients stimulated with PUREGON
Two discrete cells | 26-28 hours after fertilization
  The first observation of two discrete cells in embryos of patients stimulated with ELONVA versus embryos of patients stimulated with PUREGON
Three discrete cells | 28-44 hours after fertilization
  The first observation of three discrete cells in embryos of patients stimulated with ELONVA versus embryos of patients stimulated with PUREGON
Four discrete cells | 44-45 hours after fertilization
  The first observation of four discrete cells in embryos of patients stimulated with ELONVA versus embryos of patients stimulated with PUREGON
Five discrete cells | 44-68 hours after fertilization
  The first observation of five discrete cells in embryos of patients stimulated with ELONVA versus embryos of patients stimulated with PUREGON
Six discrete cells | 44-68 hours after fertilization
  The first observation of six discrete cells in embryos of patients stimulated with ELONVA versus embryos of patients stimulated with PUREGON
Seven discrete cells | 44-68 hours after fertilization
  The first observation of seven discrete cells in embryos of patients stimulated with ELONVA versus embryos of patients stimulated with PUREGON
Eight discrete cells | 68-69 hours after fertilization
  The first observation of eight discrete cells in embryos of patients stimulated with ELONVA versus embryos of patients stimulated with PUREGON
Nine discrete cells | 69-92 hours after fertilization
  The first observation of nine discrete cells in embryos of patients stimulated with ELONVA versus embryos of patients stimulated with PUREGON
Morula stage | 92 hours after fertilization
  End of the compaction process; when observable compaction is complete in embryos of patients stimulated with ELONVA versus embryos of patients stimulated with PUREGON

SECONDARY OUTCOMES:
Number of oocytes retrieved | Number of oocytes retrieved will be evaluated after one treatment cycle (each cycle is between 28 and 35 days)
  The influence of ELONVA versus PUREGON on the number of oocytes retrieved will be assessed.
Stage of oocyte development | Stage of oocytes retrieved will be evaluated after one treatment cycle (each cycle is between 28 and 35 days)
  The influence of ELONVA versus PUREGON on the maturity stage of oocytes (germinal vesicle, metaphase I (MI) or MII phase) retrieved will be assessed.
Fertilized oocytes | Number of fertilized oocytes will be evaluated after one treatment cycle (each cycle is between 28 and 35 days)
  The influence of ELONVA versus PUREGON on the number of fertilized oocytes will be assessed.
Embryo grading | The quality of embryos will be evaluated after one treatment cycle (each cycle is between 28 and 35 days)
  The influence of ELONVA versus PUREGON on embryo grading (Istanbul consensus criteria) will be assessed. The grading consists of assessment of cell number, fragmentation, multinucleation, cell size, cytoplasmic granularity, membrane appearance, and the presence of vacuoles).
Biochemical pregnancy (measurement of beta hCG) | Biochemical pregnancies will be evaluated after successful implantation (1 week after embryo transfer)
  The influence of Elonva versus Puregon on the number of biochemical pregnancies will be assessed.
Life birth | Life births will be evaluated after successful pregnancy (9 moths after embryo transfer)
  The influence of Elonva versus Puregon on the number of life births will be assessed.
Weight (kilograms) | Weight of the newborn will be evaluated after birth (9 moths after embryo transfer)
  The influence of Elonva versus Puregon on the weight of the newborn will be assessed.
Height (centimeters) | Height of the newborn will be evaluated after birth (9 moths after embryo transfer)
  The influence of Elonva versus Puregon on the height of the newborn will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schenk, Dr., Principal Investigator — Das Kinderwunsch Institut Schenkg GmbH
Locations (1):
- Das Kinderwunsch Institut Schenk GmbH, Dobl, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided
It has to be clarified with MERCK if sharing of data is applicable for this project.

REFERENCES:
- [Background] Gryshchenko MG, Pravdyuk AI, Parashchyuk VY. Analysis of factors influencing morphokinetic characteristics of embryos in ART cycles. Gynecol Endocrinol. 2014 Oct;30 Suppl 1:6-8. doi: 10.3109/09513590.2014.945763. PMID 25200818
- [Background] Wissing ML, Bjerge MR, Olesen AI, Hoest T, Mikkelsen AL. Impact of PCOS on early embryo cleavage kinetics. Reprod Biomed Online. 2014 Apr;28(4):508-14. doi: 10.1016/j.rbmo.2013.11.017. Epub 2013 Dec 17. PMID 24581983
- [Background] Chawla M, Fakih M, Shunnar A, Bayram A, Hellani A, Perumal V, Divakaran J, Budak E. Morphokinetic analysis of cleavage stage embryos and its relationship to aneuploidy in a retrospective time-lapse imaging study. J Assist Reprod Genet. 2015 Jan;32(1):69-75. doi: 10.1007/s10815-014-0372-3. Epub 2014 Nov 14. PMID 25395178
- [Background] Armstrong S, Vail A, Mastenbroek S, Jordan V, Farquhar C. Time-lapse in the IVF-lab: how should we assess potential benefit? Hum Reprod. 2015 Jan;30(1):3-8. doi: 10.1093/humrep/deu250. Epub 2014 Oct 14. PMID 25316446
- [Background] Milewski R, Kuc P, Kuczynska A, Stankiewicz B, Lukaszuk K, Kuczynski W. A predictive model for blastocyst formation based on morphokinetic parameters in time-lapse monitoring of embryo development. J Assist Reprod Genet. 2015 Apr;32(4):571-9. doi: 10.1007/s10815-015-0440-3. Epub 2015 Feb 18. PMID 25690157
- [Background] VerMilyea MD, Tan L, Anthony JT, Conaghan J, Ivani K, Gvakharia M, Boostanfar R, Baker VL, Suraj V, Chen AA, Mainigi M, Coutifaris C, Shen S. Computer-automated time-lapse analysis results correlate with embryo implantation and clinical pregnancy: a blinded, multi-centre study. Reprod Biomed Online. 2014 Dec;29(6):729-36. doi: 10.1016/j.rbmo.2014.09.005. Epub 2014 Sep 21. PMID 25444507